CLINICAL TRIAL: NCT05365035
Title: A Phase II Study of Cladribine and Low Dose Cytarabine in Combination With Venetoclax, Alternating With Azacitidine and Venetoclax, in Patients With Higher-risk Myeloproliferative Chronic Myelomonocytic Leukemia or Higher-risk Myelodysplastic Syndromes With Excess Blasts
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1116; NCI-2022-03803 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-04-26; First posted 2022-05-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndromes; Myeloproliferative Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Cladribine; Cytarabine; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- cladribine, cytarabine, venetoclax, and azacitidine (Experimental): Participants will receive cladribine, cytarabine, and venetoclax for 2 cycles and then azacitidine and venetoclax for 2 cycles. Participants will repeat this pattern of 2 cycles each for up to a total of 18
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Cladribine — Given by Vein (IV)
  Other Names: Leustatin®; 2-CdA
Drug: Cytarabine — Given under the skin; subcutaneous injection (SQ)
  Other Names: Ara-C; Cytosar®; DepoCyt™; Cytosine arabinosine hydrochloride
Drug: Venetoclax — Given by PO
  Other Names: ABT-199; GDC-0199
Drug: Azacitidine — Given by IV or subcutaneous injection (SQ)
  Other Names: 5-azacytidine; 5-aza; Vidaza™; 5-AZC; AZA-CR; Ladakamycin

SUMMARY:
To learn if the combination of cladribine, cytarabine, venetoclax, and azacitidine can help to control higher-risk myelodysplastic syndrome (MDS) with excess blasts and/or higher-risk chronic myelomonocytic leukemia (CMML).

DETAILED DESCRIPTION:
Primary Objectives:

* To determine the efficacy, safety and tolerability of the combination of cladribine, cytarabine and venetoclax in higher-risk MDS with excess blasts and higher-risk CMML.
* MDS relapsed cohort (Cohort A, N=20): MDS with Int-2 or High risk IPSS and >5% blasts with no response after 6 cycles of azacitidine, decitabine, guadecitabine, CC-486 or ASTX727 (decitabine/cedazuridine) or relapse or progression after any number of cycles
* CMML relapsed cohort (Cohort B, N=10): CMML 1 or 2 with no response after 6 cycles of azacitidine, decitabine, guadecitabine, CC-486 or ASTX727 (decitabine/cedazuridine) or relapse or progression after any number of cycles
* MDS HMA-naïve cohort (Cohort C, N=20): MDS with Int-2 or High risk by IPSS and >10% blasts OR diagnosis
* CMML HMA-naïve cohort (Cohort D, N=10): CMML-2; OR CMML-1 with at least one of the following high-risk features: extramedullary disease, splenomegaly of >5cm below costal margin, platelets <100x109/L, Hgb level <10g/dL, WBC >13x109/L, clonal cytogenetic abnormality (other than monosomy Y).

Secondary Objectives:

* To evaluate responses by 2015 IWG MDS/MPN response criteria in patients with MDS/MPN and by 2023 IWG response criteria in all patients (Appendix).
* To assess overall survival (OS), duration of response, leukemia-free survival (LFS), and relapse-free survival (RFS).
* To evaluate proportion of transplant-candidate patients bridged to allogeneic stem-cell transplant.
* Correlative studies including correlation of response with disease subtype and genomic profile.
* To evaluate changes in clonal composition and VAF of identified mutations with therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years.
2. Diagnosis of MDS or CMML by WHO and:

   * MDS relapsed cohort (Cohort A): MDS with IPSS-R score >3.5 and >5% blasts with no response after 6 cycles of azacitidine, decitabine, guadecitabine or ASTX727 (decitabine/cedazuridine) or relapse or progression after any number of cycles
   * CMML relapsed cohort (Cohort B): CMML 1 or 2 with no response after 6 cycles of azacitidine, decitabine, guadecitabine or ASTX727 (decitabine/cedazuridine) or relapse or progression after any number of cycles
   * MDS HMA-naïve cohort (Cohort C): MDS with IPSS-R score >3.5 and >/= 10% blasts
   * CMML HMA-naïve cohort (Cohort D): CMML-2; OR CMML-1 with at least one of the following high-risk features: extramedullary disease, splenomegaly of >5cm below costal margin or by sonographic volumetric assessment, platelets <100x109/L, Hgb level <10g/dL, WBC >13x109/L, clonal cytogenetic abnormality (other than monosomy Y) or high risk mutations (ASXL1, RUNX1, SETBP1, BRAF, NRAS, KRAS, PTPN11, NF1, CBL).
   * MDS/MPN relapsed cohort (Cohort E): MDS/MPN-NOS, MDS/MPN with neutrophilia (atypical CML) or MDS/MPN-RS-T with >5% blasts with no response after 6 cycles of azacitidine, decitabine, guadecitabine or ASTX727 (decitabine/cedazuridine) or relapse or progression after any number of cycles
   * MDS/MPN HMA-naïve cohort (Cohort F): MDS/MPN-NOS or MDS/MPN with neutrophilia (atypical CML) with

     * >/=10% blasts or
     * with >5% blasts at least one of the following high-risk features: splenomegaly >5cm below costal margin, WBC >13x109/L, high risk cytogenetic or molecular features (ASXL1, SETBP1, i(17q), TP53) or
     * who might not be deemed to benefit from HMA therapy due to proliferative or extramedullary disease.
3. Eastern Cooperative Oncology Group (ECOG) performance status of </= 2
4. Creatinine clearance > 30 ml/min no end/stage renal disease (using Cockcroft-Gault)
5. Adequate hepatic function with total bilirubin 2x ULN, AST or ALT 2.5 xULN unless deemed to be due to underlying disease involvement.
6. Willing to adhere to and comply with all prohibitions and restrictions specified in the protocol.
7. Patient must have signed an informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study.
8. English and Non-English speaking patients will be allowed

Exclusion Criteria:

1. Uncontrolled infection not adequately responding to appropriate antibiotics
2. New York Heart Association (NYHA) Class III or IV congestive heart failure or LVEF <50% by echocardiogram or multigated acquisition (MUGA) scan.
3. History of myocardial infarction within the last 6 months or unstable/uncontrolled angina pectoris or history of severe and/or uncontrolled ventricular arrhythmias.
4. Female patients who are pregnant or lactating.
5. Patients with reproductive potential who are unwilling to following contraception requirements (including condom use for males with sexual partners, and for females: prescription oral contraceptives [birth control pills], contraceptive injections, intrauterine devices [IUD], double-barrier method [spermidical jelly or foam with condoms or diaphragm], contraceptive patch, or surgical sterilization) throughout the study.
6. Female patients with reproductive potential who do not have a negative urine or blood beta-human chorionic gonadotropin (beta HCG) pregnancy test at screening.
7. Patients receiving any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish the overall survival (OS). | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Bravo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT05365035/ICF_000.pdf